CLINICAL TRIAL: NCT02283190
Title: 1336GCC: Open-Label, Single-Arm PK Study of IV Erwinaze (Asparaginase Erwinia Chrysanthemi) to Find the Dose With Acceptable Therapeutic and Safety Profile in Adults With Acute Myeloid Leukemia With or Without Isocitrate Dehydrogenase Mutations
Brief Title: 1336GCC: Study of Erwinaze for Treatment of Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ashkan Emadi (Other)
Responsible Party: Sponsor-Investigator, Ashkan Emadi, Sponsor-Investigator, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1336GCC, HP-00056335
Record Dates: First submitted 2014-10-17; First posted 2014-11-05 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Asparaginase; Glutamine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Asparaginase; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ewwinase (Experimental): Six doses of Erwinase given three times weekly (Monday-Wednesday-Friday) for two weeks. Possible dose levels used are 20.000 IU/m2/day, 25,000IU/m2/day, and 30,000IU/m2/day.
  Interventions: Drug: Erwinase

INTERVENTIONS:
Drug: Erwinase — Six doses of Erwinase, given Monday-Wednesday-Friday for 2 weeks. Dosage levels to be used are: 20,000 IU/ m2 /day, 25,000 IU/ m2 /day, 30,000 IU/ m2 /day.
  Other Names: Asparaginase; Crisantaspase

SUMMARY:
Erwinaze will be administered intravenously at a dose of 25,000 IU/m2 (dose cohort 0) for 6 doses MWF over a period of 2 weeks to 9 patients (as described below and in the following schema). Blood counts, chemistries including bilirubin, amylase and lipase, and coagulation studies including fibrinogen will be measured and reviewed before each asparaginase dose. Fibrinogen (<100 mg/dL) can be replaced with cryoprecipitate before each dose at the discretion of treating physician. Treatment will be stopped for elevation of amylase, lipase or direct bilirubin above normal range.

DETAILED DESCRIPTION:
For safety:

Erwinaze has been already used in clinical practice for treatment of patients with acute leukemia with known side effect profile. For this reason, in this protocol, we use the "3+3+3" design for evaluation of safety based on pre-determined dose-limiting toxicities (DLT). In the "3+3+3" design, the dose escalation rules proceed by adjusting the dose in cohorts of 3 to 9 patients per three dose levels:20,000 IU/m2 (dose cohort -1), 25,000 IU/m2 (dose cohort 0), 30,000 IU/m2 (dose cohort +1). The goal is to determine the Recommended Phase 2 Dose (RP2D)

For anti-leukemic activity:

To evaluate the activity of Erwinaze to reduce the serum glutamine to the desired level, the dose will be adjusted according to a pre-defined algorithm based on 48-hour trough serum glutamine level (biochemical response) prior to dose 6 of each patient. If the safety profile is acceptable, we will enroll up to a total of 15 patients at that dose level to better study and analyze the glutamine-reducing effect of Erwinaze at the defined dose.

In summary, if 9 patients are treated at a certain dose and at least 7 out of 9 individuals respond to treatment (per serum glutamine levels) and < 3 develop DLT, this dose level will be declared the Recommended Phase 2 Dose (RP2D). Six additional patients (total of 15 to 18 patients) will be enrolled at the RP2D level to better assess toxicity and to document responses.

There will be no intra-patient dose escalation or reduction.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed AML
* 18 years and older
* AML has relapsed after, or is refractory to, first-line therapy, with or without subsequent additional therapy
* Have received or are ineligible for immediate established curative regimens
* ASCT patients are eligible provided that they are >= 4 weeks from stem cell infusion
* alloSCT patients are eligible if they are >= 60 days post stem cell infusion, have no evidence of graft versus host disease (GVHD) > Grade 1, and are >= 2 weeks off all immunosuppressive therapy
* Previous cytotoxic chemotherapy completed at least 3 weeks and radiotherapy at least 2 weeks prior to day 1 of study treatment
* Biologic agents stopped at least 1 week prior to day 1 of study treatment
* DNA methyltransferase inhibitors stopped at least 3 weeks prior to day 1 of study treatment
* ECOG performance status ≤2
* Patients must have normal organ function
* Female patients of childbearing potential must have a negative pregnancy test.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving any other investigational agents, or concurrent chemotherapy, radiation therapy, or immunotherapy
* Patients with acute promyelocytic leukemia
* Patients with active central nervous system leukemia
* Prior treatment with Erwinaze
* Hyperleukocytosis with > 50,000 blasts/μL
* History of a major thrombotic event
* History of pancreatitis
* Active, uncontrolled infection
* Uncontrolled intercurrent illness
* Pregnant women
* Uncontrolled active seizure disorder or a history of seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To determine the dose of Erwinase that produces a plasma glutamine level ≤120 μmol/L with an acceptable safety profile. | Day 3
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.
Efficacy of Erwinase doses as measured by plasma glutamine level | Day 5
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.
Efficacy of Erwinase doses as measured by plasma glutamine level | Day 8
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.
Efficacy of Erwinase doses as measured by plasma glutamine level | Day 10
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.
Efficacy of Erwinase doses as measured by plasma glutamine level | Day 12
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.
Efficacy of Erwinase doses as measured by plasma glutamine level | Day 42
  The dose of Erwinase that produces a plasma glutamine level ≤120 µmol/L with an acceptable safety profile.

SECONDARY OUTCOMES:
Efficacy of Erwinase doses as measured by nadir serum asparaginase activity | Days 3, 5,8,10,12, & 42
  The dose of Erwinase that produces nadir serum asparaginase activity ≥0.1 IU/mL with acceptable safety profile.
Efficacy of Erwinase as measured by acute myeloid leukemia (AML) disease response | Days 15 and 29
  Bone marrow biopsy to determine the clinical response to 6 doses of Erwinaze at the administered dose.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days from last dose of drug or until death, whichever occurs first
  To establish safety and tolerability of Erwinaze in patients with AML with or without mIDH
Validity of serum and urine 2-hydroxyglutarate (2-HG) as a biomarker for AML with or without IDH mutation | Days 0, 8, & 42
  Measure the blood and urine 2-hydroxyglutarate (2-HG) levels

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Emadi, MD, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States